CLINICAL TRIAL: NCT06632041
Title: Haematological Disturbances in Neonates with Necrotizing Enterocolities
Brief Title: Necrotizing Enterocolities
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mervat maher saad zakhary, Principal investigator, Assiut University
Other Study IDs: Necrotizing enterocolities
Record Dates: First submitted 2024-10-06; First posted 2024-10-08 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Necrotizing Enterocolitis of Newborn
MeSH Terms: interventions — Blood Cell Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Neonates with necrotizing enterocolities
  Interventions: Diagnostic Test: Complete blood count; Other: Complete blood count

INTERVENTIONS:
Diagnostic Test: Complete blood count — Study haemtological disturbances in neonates with necrotizing enterocolities
Other: Complete blood count — Haemtological disturbances in neonates with necrotizing enterocolities

SUMMARY:
Haematological disturbances in neonates with necrotizing enterocolities

DETAILED DESCRIPTION:
Necrotizing enterocolitis (NEC) is an acquired, multifactorial and devastating gastrointestinal disease associated with high morbidity and mortality in preterm neonates. With an incidence of about 7% in infants with BW < 1500 g and mortality up to 30%, NEC presents as a medical and surgical emergency It is characterized by ischemia, necrosis, and inflammation of bowel wall with invasion by gas-forming organisms and intramural dissection of gas ,characteristicall appearing as pneumatosis intestinalis in radiological and pathological studies. While exact etiology is undetermined, the pathogenesis is believed to be an anomalous innate immune response to an altered, less diverse intestinal microbiota by the highly immunoreactive enterocytes of premature infants, leading to inflammation and tissue necrosis

* in this devastating disease with undetermined etiology. Breast milk feeding, prolonging gestation to avoid prematurity, antenatal steroid, and the use of probiotics/prebiotics are established prevention strategies in NEC
* The hematological abnormalities associated with NEC were first described 25 years ago by Hutter et al.The abnormalities observed in a series of 40 patients with NEC included thrombocytopenia, with
* and without disseminated intravascular coagulation (DIC), neutrophilia or neutropenia, and hemolytic anemia.

ELIGIBILITY:
Inclusion Criteria:

* preterm less than 36 weeks
* Or very low birth weight less than 1500 gram

Exclusion Criteria:

* full term
* Normal birth weight ,Preterm with early breast feeding or more than 1500 gm

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates with necrotizing enterocolities
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Aim | Baseline
  :to delineate haemtological abnormalities in neonatal necrotizing enterocolities as predictors of morbidity and mortality